CLINICAL TRIAL: NCT02638103
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group Study Evaluating the Long-Term Safety, Tolerability, and Efficacy of Subcutaneous Administration of Fremanezumab (TEV-48125) for the Preventive Treatment of Migraine
Brief Title: Efficacy and Safety of Subcutaneous Administration of Fremanezumab (TEV-48125) for the Preventive Treatment of Migraine
Acronym: HALO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV48125-CNS-30051; 2015-004550-18 (EudraCT Number)
Expanded Access: NCT03539393 (Available)
Record Dates: First submitted 2015-12-18; First posted 2015-12-22 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — fremanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TEV-48125 225 mg Monthly: New/Placebo Rollover Participants (Experimental): Participants with CM who were randomized to the placebo treatment group or participants who do not rollover from the pivotal efficacy study, will receive fremanezumab 675 milligrams (mg) SC as loading dose (3 injections of fremanezumab 225 mg/1.5 milliliters [mL] on Day 0) followed by 11 monthly SC doses of fremanezumab at 225 mg (1 injection of fremanezumab 225 mg/1.5 mL and 2 injections of placebo 1.5 mL on Days 84, 168, and 252; and 1 injection of fremanezumab 225 mg/1.5mL on Days 28, 56, 112, 140, 196, 224, 280, and 308). Participants with EM who were randomized to the placebo treatment group or participants who do not rollover from the pivotal efficacy study, will receive 12 monthly SC doses of fremanezumab at 225 mg (1 injection of fremanezumab 225 mg/1.5 mL and 2 injections of placebo 1.5 mL on Days 0, 84, 168, and 252; and 1 injection of fremanezumab 225 mg/1.5 mL on Days 28, 56, 112, 140, 196, 224, 280, and 308).
  Interventions: Drug: Fremanezumab; Drug: Placebo
- TEV-48125 225 mg Monthly: Active Rollover Participants (Experimental): Participants with CM who were randomized to the active treatment group (Fremanezumab 675/225 mg) in the pivotal efficacy study, will receive fremanezumab 675 mg SC as loading dose (3 injections of fremanezumab 225 mg/1.5 mL on Day 0) followed by 11 monthly SC doses of fremanezumab at 225 mg (1 injection of fremanezumab 225 mg/1.5mL and 2 injections of placebo 1.5 mL on Days 84, 168, and 252; and 1 injection of fremanezumab 225 mg/1.5mL on Days 28, 56, 112, 140, 196, 224, 280, and 308). Participants with EM who were randomized to the active treatment group (Fremanezumab 225 mg) in the pivotal efficacy study, will receive 12 monthly SC doses of fremanezumab at 225 mg (1 injection of fremanezumab 225 mg/1.5 mL and 2 injections of placebo 1.5 mL on Days 0, 84, 168, and 252; and 1 injection of fremanezumab 225 mg/1.5 mL on Days 28, 56, 112, 140, 196, 224, 280, and 308).
  Interventions: Drug: Fremanezumab; Drug: Placebo
- TEV-48125 675 mg Quarterly: New/Placebo Rollover Participants (Experimental): Participants with CM or EM who were randomized to the placebo treatment group or participants who do not rollover from the pivotal efficacy study, will receive fremanezumab 675 mg SC once every 3 months for 12 months for a total of 4 doses (3 injections of fremanezumab 225 mg/1.5 mL on Days 0, 84, 168, and 252; and 1 injection of placebo 1.5 mL on Days 28, 56, 112, 140, 196, 224, 280, and 308).
  Interventions: Drug: Fremanezumab; Drug: Placebo
- TEV-48125 675 mg Quarterly: Active Rollover Participants (Experimental): Participants with CM or EM who were randomized to the active treatment group (Fremanezumab 675 mg) in the pivotal efficacy study, will receive fremanezumab 675 mg SC once every 3 months for 12 months for a total of 4 doses (3 injections of fremanezumab 225 mg/1.5 mL on Days 0, 84, 168, and 252; and 1 injection of placebo 1.5 mL on Days 28, 56, 112, 140, 196, 224, 280, and 308).
  Interventions: Drug: Fremanezumab; Drug: Placebo

INTERVENTIONS:
Drug: Fremanezumab — Fremanezumab will be administered as per the dose and schedule specified in the respective arms.
  Other Names: TEV-48125
Drug: Placebo — Placebo matching to fremanezumab will be administered as per schedule specified in the respective arms.

SUMMARY:
A study to evaluate the long-term safety, tolerability, and efficacy of subcutaneous (SC) administration of TEV-48125 in adult participants with chronic migraine (CM) or episodic migraine (EM). Participants with CM or EM who complete the pivotal efficacy studies of TEV-48125 (TV48125-CNS-30049 [NCT02621931] and TV48125-CNS-30050 [NCT02629861]) and agree to participate in this study; and new participants meeting eligibility criteria (not rolling over from pivotal studies), will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

Participants Rolling Over from the Pivotal Efficacy Studies:

* Participant must have signed and dated the informed consent document.
* Participant must have completed the pivotal efficacy study without major protocol violations.

  * Additional criteria apply, please contact the investigator for more information.

Participants Not Rolling Over from the Pivotal Efficacy Studies:

* Males or females aged 18 to 70 years, inclusive, with migraine onset at less than or equal to (≤) 50 years of age.
* Participant signed and dated the informed consent document.
* Participant has a history of migraine or clinical judgment suggests a migraine diagnosis.
* Participant fulfills the criteria for EM or CM with prospectively collected baseline information during the 28-day run-in period.
* Body mass index (BMI) of 17.5 to 37.5 kilograms/square meter (kg/m^2) and a total body weight between 45 and 120 kg, inclusive.
* All participants must be of non-childbearing potential.

  1. Participants must simultaneously use 2 forms of highly effective contraception methods.
  2. Participants will remain abstinent throughout the study.
* Female participants of childbearing potential must have a negative serum beta-human chorionic gonadotropin (β-HCG) pregnancy test prior at screening (confirmed by urine dipstick β-HCG pregnancy test at baseline).
* The participant must be willing and able to comply with study restrictions, to remain at the clinic for the required duration during the study period, and to return to the clinic for the follow-up evaluation.

  * Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

Participants Rolling Over from the Pivotal Efficacy Studies:

* Pregnant or nursing females
* Compliance with daily diary entry lower than 75 percent (%) at the last month of the double-blind treatment period of the pivotal efficacy study.

  * Additional criteria apply, please contact the investigator for more information.

Participants Not Rolling Over from the Pivotal Efficacy Studies:

* Clinically significant findings at the discretion of the investigator.
* Evidence or medical history of clinically significant psychiatric issues, including any suicide attempt in the past, or suicidal ideation with a specific plan in the past 2 years.
* History of clinically significant cardiovascular disease or vascular ischemia (such as myocardial, neurological [for example; cerebral ischemia], peripheral extremity ischemia, or other ischemic event) or thromboembolic events (arterial or venous thrombotic or embolic events) such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism -Known infection or history of human immunodeficiency virus, tuberculosis, or chronic hepatitis B or C infection.
* Past or current history of cancer in the past 5 years, except for appropriately treated nonmelanoma skin carcinoma.
* Pregnant or nursing females.
* History of hypersensitivity reactions to injected proteins, including monoclonal antibodies.
* Participation in a clinical study of a new chemical entity or a prescription medicine within 2 months before study drug administration or 5 half-lives, whichever is longer.
* History of alcohol or drug abuse during the past 2 years, or alcohol or drug dependence during the past 5 years.
* The participant cannot participate or successfully complete the study, in the opinion of their healthcare provider or the investigator, for any of the following reasons:

  1. mentally or legally incapacitated or unable to give consent for any reason.
  2. in custody due to an administrative or a legal decision, under guardianship, or institutionalized.
  3. unable to be contacted in case of emergency.
  4. has any other condition, which, in the opinion of the investigator, makes the participant inappropriate for inclusion in the study.
* Participant is a study center or sponsor employee who is directly involved in the study or the relative of such an employee.

  * Additional criteria apply, please contact the investigator for more information.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1890 (Actual)
Dates: Start 2016-02-26 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (139):
- United States (90):
  - Teva Investigational Site 13628, Birmingham, Alabama
  - Teva Investigational Site 13577, Birmingham, Alabama
  - Teva Investigational Site 13606, Phoenix, Arizona
  - Teva Investigational Site 13579, Phoenix, Arizona
  - Teva Investigational Site 13602, Little Rock, Arkansas
  - Teva Investigational Site 13568, Encino, California
  - Teva Investigational Site 13546, Fullerton, California
  - Teva Investigational Site 13540, Long Beach, California
  - Teva Investigational Site 13632, Redlands, California
  - Teva Investigational Site 13571, Redondo Beach, California
  - Teva Investigational Site 13573, San Diego, California
  - Teva Investigational Site 13538, Santa Monica, California
  - Teva Investigational Site 13594, Santa Rosa, California
  - Teva Investigational Site 13595, Walnut Creek, California
  - Teva Investigational Site 13629, Aurora, Colorado
  - Teva Investigational Site 13557, Boulder, Colorado
  - Teva Investigational Site 13593, Colorado Springs, Colorado
  - Teva Investigational Site 13633, Denver, Colorado
  - Teva Investigational Site 13612, Denver, Colorado
  - Teva Investigational Site 13631, Englewood, Colorado
  - Teva Investigational Site 13563, East Hartford, Connecticut
  - Teva Investigational Site 13550, Stamford, Connecticut
  - Teva Investigational Site 13635, Bradenton, Florida
  - Teva Investigational Site 13597, Gainesville, Florida
  - Teva Investigational Site 13607, Hialeah, Florida
  - Teva Investigational Site 13559, Jacksonville, Florida
  - Teva Investigational Site 13584, Ocala, Florida
  - Teva Investigational Site 13587, Orlando, Florida
  - Teva Investigational Site 13567, Palm Beach Gardens, Florida
  - Teva Investigational Site 13553, Pembroke Pines, Florida
  - Teva Investigational Site 13616, Pinellas Park, Florida
  - Teva Investigational Site 13620, Atlanta, Georgia
  - Teva Investigational Site 13537, Atlanta, Georgia
  - Teva Investigational Site 13604, Boise, Idaho
  - Teva Investigational Site 13585, Chicago, Illinois
  - Teva Investigational Site 13621, Chicago, Illinois
  - Teva Investigational Site 13627, Evanston, Illinois
  - Teva Investigational Site 13596, Indianapolis, Indiana
  - Teva Investigational Site 13617, Wichita, Kansas
  - Teva Investigational Site 13598, Wichita, Kansas
  - Teva Investigational Site 13566, Louisville, Kentucky
  - Teva Investigational Site 13603, Metairie, Louisiana
  - Teva Investigational Site 13582, Pikesville, Maryland
  - Teva Investigational Site 13590, Boston, Massachusetts
  - Teva Investigational Site 13589, New Bedford, Massachusetts
  - Teva Investigational Site 13543, Watertown, Massachusetts
  - Teva Investigational Site 13539, Ann Arbor, Michigan
  - Teva Investigational Site 13542, Golden Valley, Minnesota
  - Teva Investigational Site 13534, Kansas City, Missouri
  - Teva Investigational Site 13536, Springfield, Missouri
  - Teva Investigational Site 13619, St Louis, Missouri
  - Teva Investigational Site 13618, Fremont, Nebraska
  - Teva Investigational Site 13605, Las Vegas, Nevada
  - Teva Investigational Site 13578, Lebanon, New Hampshire
  - Teva Investigational Site 13575, Martinsville, New Jersey
  - Teva Investigational Site 13622, Princeton, New Jersey
  - Teva Investigational Site 13588, Albuquerque, New Mexico
  - Teva Investigational Site 13576, Amherst, New York
  - Teva Investigational Site 13565, Plainview, New York
  - Teva Investigational Site 13544, Greensboro, North Carolina
  - Teva Investigational Site 13574, Greensboro, North Carolina
  - Teva Investigational Site 13545, Raleigh, North Carolina
  - Teva Investigational Site 13609, Akron, Ohio
  - Teva Investigational Site 13625, Akron, Ohio
  - Teva Investigational Site 13634, Akron, Ohio
  - Teva Investigational Site 13533, Cincinnati, Ohio
  - Teva Investigational Site 13624, Cincinnati, Ohio
  - Teva Investigational Site 13569, Cleveland, Ohio
  - Teva Investigational Site 13626, Columbus, Ohio
  - Teva Investigational Site 13561, Oklahoma City, Oklahoma
  - Teva Investigational Site 13601, Eugene, Oregon
  - Teva Investigational Site 13591, Jenkintown, Pennsylvania
  - Teva Investigational Site 13554, Philadelphia, Pennsylvania
  - Teva Investigational Site 13608, Uniontown, Pennsylvania
  - Teva Investigational Site 13615, Greer, South Carolina
  - Teva Investigational Site 13556, Mt. Pleasant, South Carolina
  - Teva Investigational Site 13560, Bristol, Tennessee
  - Teva Investigational Site 13551, Memphis, Tennessee
  - Teva Investigational Site 13532, Nashville, Tennessee
  - Teva Investigational Site 13552, Nashville, Tennessee
  - Teva Investigational Site 13541, Austin, Texas
  - Teva Investigational Site 13623, Dallas, Texas
  - Teva Investigational Site 13611, Plano, Texas
  - Teva Investigational Site 13572, San Antonio, Texas
  - Teva Investigational Site 13614, Murray, Utah
  - Teva Investigational Site 13581, West Jordan, Utah
  - Teva Investigational Site 13630, Virginia Beach, Virginia
  - Teva Investigational Site 13564, Seattle, Washington
  - Teva Investigational Site 13586, Seattle, Washington
  - Teva Investigational Site 13600, Morgantown, West Virginia
- Canada (5):
  - Teva Investigational Site 11124, Hamilton, Ontario
  - Teva Investigational Site 11122, Newmarket, Ontario
  - Teva Investigational Site 11120, Calgary
  - Teva Investigational Site 11121, Montreal
  - Teva Investigational Site 11123, Sarnia
- Czechia (6):
  - Teva Investigational Site 54144, Brno
  - Teva Investigational Site 54141, Kunratice
  - Teva Investigational Site 54145, Pardubice
  - Teva Investigational Site 54143, Prague
  - Teva Investigational Site 54146, Prague
  - Teva Investigational Site 54142, Prague
- Finland (3):
  - Teva Investigational Site 40018, Helsinki
  - Teva Investigational Site 40017, Helsinki
  - Teva Investigational Site 40016, Turku
- Israel (6):
  - Teva Investigational Site 80096, Holon
  - Teva Investigational Site 80099, Jerusalem
  - Teva Investigational Site 80098, Nahariya
  - Teva Investigational Site 80097, Netanya
  - Teva Investigational Site 80100, Ramat Gan
  - Teva Investigational Site 80095, Tel Aviv
- Japan (13):
  - Teva Investigational Site 84072, Chofu-shi
  - Teva Investigational Site 84066, Kagoshima
  - Teva Investigational Site 84069, Kai
  - Teva Investigational Site 84073, Kawasaki
  - Teva Investigational Site 84067, Kyoto
  - Teva Investigational Site 84062, Osaka
  - Teva Investigational Site 84070, Saitama
  - Teva Investigational Site 84061, Sendai
  - Teva Investigational Site 84063, Shinjuku-ku
  - Teva Investigational Site 84068, Shizuoka
  - Teva Investigational Site 84065, Tochigi
  - Teva Investigational Site 84064, Tokyo
  - Teva Investigational Site 84071, Toyonaka
- Poland (5):
  - Teva Investigational Site 53364, Krakow
  - Teva Investigational Site 53363, Krakow
  - Teva Investigational Site 53366, Lublin
  - Teva Investigational Site 53365, Poznan
  - Teva Investigational Site 53367, Warsaw
- Russia (7):
  - Teva Investigational Site 50399, Kazan'
  - Teva Investigational Site 50395, Kazan'
  - Teva Investigational Site 50394, Moscow
  - Teva Investigational Site 50400, Moscow
  - Teva Investigational Site 50398, Nizhny Novgorod
  - Teva Investigational Site 50396, Nizhny Novgorod
  - Teva Investigational Site 50397, Ufa
- Spain (4):
  - Teva Investigational Site 31207, Madrid
  - Teva Investigational Site 31208, Pamplona
  - Teva Investigational Site 31205, Valladolid
  - Teva Investigational Site 31206, Zaragoza

REFERENCES:
- [Derived] Goadsby PJ, Silberstein SD, Yeung PP, Cohen JM, Ning X, Yang R, Dodick DW. Long-term safety, tolerability, and efficacy of fremanezumab in migraine: A randomized study. Neurology. 2020 Nov 3;95(18):e2487-e2499. doi: 10.1212/WNL.0000000000010600. Epub 2020 Sep 10. PMID 32913018
- [Derived] Buse DC, Gandhi SK, Cohen JM, Ramirez-Campos V, Cloud B, Yang R, Cowan RP. Improvements across a range of patient-reported domains with fremanezumab treatment: results from a patient survey study. J Headache Pain. 2020 Sep 4;21(1):109. doi: 10.1186/s10194-020-01177-4. PMID 32887548

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with chronic or episodic migraine (CM or EM) who completed the pivotal efficacy studies of fremanezumab (TV48125-CNS-30049 [NCT02621931] and TV48125-CNS-30050 [NCT02629861]) and agreed to participate in this study; and new participants meeting eligibility criteria (not rolling over from pivotal studies), were enrolled in this study.
Pre-assignment Details: A total of 1890 participants were enrolled, including 917 participants with CM rolled over from Study TV48125-CNS-30049, 661 participants with EM rolled over from Study TV48125-CNS-30050, and 312 newly enrolled participants (193 with CM and 119 with EM).
Groups:
- TEV-48125 225 mg Monthly: New/Placebo Rollover Participants: Participants with CM who were randomized to the placebo treatment group or participants who did not rollover from the pivotal efficacy study, received fremanezumab (TEV-48125) 675 milligrams (mg) subcutaneously (SC) as loading dose (3 injections of fremanezumab 225 mg/1.5 milliliters [mL] on Day 0) followed by 11 monthly SC doses of fremanezumab at 225 mg (1 injection of fremanezumab 225 mg/1.5mL and 2 injections of placebo 1.5 mL on Days 84, 168, and 252; and 1 injection of fremanezumab 225 mg/1.5mL on Days 28, 56, 112, 140, 196, 224, 280, and 308). Participants with EM who were randomized to the placebo treatment group or participants who did not rollover from the pivotal efficacy study, received 12 monthly SC doses of fremanezumab at 225 mg (1 injection of fremanezumab 225 mg/1.5 mL and 2 injections of placebo 1.5 mL on Days 0, 84, 168, and 252; and 1 injection of fremanezumab 225 mg/1.5 mL on Days 28, 56, 112, 140, 196, 224, 280, and 308).
- TEV-48125 225 mg Monthly: Active Rollover Participants: Participants with CM who were randomized to the active treatment group (Fremanezumab 675/225 mg) in the pivotal efficacy study, received fremanezumab 675 mg SC as loading dose (3 injections of fremanezumab 225 mg/1.5 mL on Day 0) followed by 11 monthly SC doses of fremanezumab at 225 mg (1 injection of fremanezumab 225 mg/1.5 mL and 2 injections of placebo 1.5 mL on Days 84, 168, and 252; and 1 injection of fremanezumab 225 mg/1.5mL on Days 28, 56, 112, 140, 196, 224, 280, and 308). Participants with EM who were randomized to the active treatment group (Fremanezumab 225 mg) in the pivotal efficacy study, received 12 monthly SC doses of fremanezumab at 225 mg (1 injection of fremanezumab 225 mg/1.5 mL and 2 injections of placebo 1.5 mL on Days 0, 84, 168, and 252; and 1 injection of fremanezumab 225 mg/1.5 mL on Days 28, 56, 112, 140, 196, 224, 280, and 308).
- TEV-48125 675 mg Quarterly: New/Placebo Rollover Participants: Participants with CM or EM who were randomized to the placebo treatment group or participants who did not rollover from the pivotal efficacy study, received fremanezumab 675 mg SC once every 3 months for 12 months for a total of 4 doses (3 injections of fremanezumab 225 mg/1.5 mL on Days 0, 84, 168, and 252; and 1 injection of placebo 1.5 mL on Days 28, 56, 112, 140, 196, 224, 280, and 308).
- TEV-48125 675 mg Quarterly: Active Rollover Participants: Participants with CM or EM who were randomized to the active treatment group (Fremanezumab 675 mg) in the pivotal efficacy study, received fremanezumab 675 mg SC once every 3 months for 12 months for a total of 4 doses (3 injections of fremanezumab 225 mg/1.5 mL on Days 0, 84, 168, and 252; and 1 injection of placebo 1.5 mL on Days 28, 56, 112, 140, 196, 224, 280, and 308).
Period: Overall Study
Arm/Group | TEV-48125 225 mg Monthly: New/Placebo Rollover Participants | TEV-48125 225 mg Monthly: Active Rollover Participants | TEV-48125 675 mg Quarterly: New/Placebo Rollover Participants | TEV-48125 675 mg Quarterly: Active Rollover Participants
Started | 419 | 526 | 420 | 525
Safety Analysis Set (Received at least 1 dose of study drug) | 418 | 526 | 419 | 525
Full Analysis Set (FAS) (Participants in safety analysis set who had at least 10 days of post-baseline efficacy assessment.) | 416 | 520 | 419 | 523
Completed | 313 | 408 | 335 | 383
Not Completed | 106 | 118 | 85 | 142
Not completed — Adverse Event | 13 | 12 | 19 | 12
Not completed — Withdrawal by Subject | 43 | 53 | 30 | 61
Not completed — Protocol Violation | 1 | 2 | 1 | 4
Not completed — Pregnancy | 2 | 3 | 0 | 1
Not completed — Non-compliance to Study Procedures | 2 | 1 | 1 | 1
Not completed — Lost to Follow-up | 26 | 33 | 20 | 37
Not completed — Lack of Efficacy | 14 | 10 | 12 | 22
Not completed — Other than specified | 5 | 4 | 2 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis set included all participants who were randomized in this study for long-term safety evaluation, regardless if they receive study treatment or not.
Groups:
- TEV-48125 225 mg Monthly: New/Placebo Rollover Participants: Participants with CM who were randomized to the placebo treatment group or participants who did not rollover from the pivotal efficacy study, received fremanezumab 675 mg SC as loading dose (3 injections of fremanezumab 225 mg/1.5 mL on Day 0) followed by 11 monthly SC doses of fremanezumab at 225 mg (1 injection of fremanezumab 225 mg/1.5 mL and 2 injections of placebo 1.5 mL on Days 84, 168, and 252; and 1 injection of fremanezumab 225 mg/1.5 mL on Days 28, 56, 112, 140, 196, 224, 280, and 308). Participants with EM who were randomized to the placebo treatment group or participants who did not rollover from the pivotal efficacy study, received 12 monthly SC doses of fremanezumab at 225 mg (1 injection of fremanezumab 225 mg/1.5 mL and 2 injections of placebo 1.5 mL on Days 0, 84, 168, and 252; and 1 injection of fremanezumab 225 mg/1.5 mL on Days 28, 56, 112, 140, 196, 224, 280, and 308).
- TEV-48125 225 mg Monthly: Active Rollover Participants: Participants with CM who were randomized to the active treatment group (Fremanezumab 675/225 mg) in the pivotal efficacy study, received fremanezumab 675 mg SC as loading dose (3 injections of fremanezumab 225 mg/1.5 mL on Day 0) followed by 11 monthly SC doses of fremanezumab at 225 mg (1 injection of fremanezumab 225 mg/1.5 mL and 2 injections of placebo 1.5 mL on Days 84, 168, and 252; and 1 injection of fremanezumab 225 mg/1.5 mL on Days 28, 56, 112, 140, 196, 224, 280, and 308). Participants with EM who were randomized to the active treatment group (Fremanezumab 225 mg) in the pivotal efficacy study, received 12 monthly SC doses of fremanezumab at 225 mg (1 injection of fremanezumab 225 mg/1.5 mL and 2 injections of placebo 1.5 mL on Days 0, 84, 168, and 252; and 1 injection of fremanezumab 225 mg/1.5 mL on Days 28, 56, 112, 140, 196, 224, 280, and 308).
- Total: Total of all reporting groups
Arm/Group | TEV-48125 225 mg Monthly: New/Placebo Rollover Participants | TEV-48125 225 mg Monthly: Active Rollover Participants | TEV-48125 675 mg Quarterly: New/Placebo Rollover Participants | TEV-48125 675 mg Quarterly: Active Rollover Participants | Total
Number analyzed (Participants) | 419 | 526 | 420 | 525 | 1890
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (12.09) | 42.9 (11.97) | 44.0 (11.67) | 43.2 (11.73) | 43.5 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 365 | 454 | 369 | 457 | 1645
  Male | 54 | 72 | 51 | 68 | 245
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 45 | 34 | 38 | 146
  Not Hispanic or Latino | 387 | 481 | 386 | 484 | 1738
  Unknown or Not Reported | 3 | 0 | 0 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 351 | 424 | 343 | 412 | 1530
  Black | 32 | 38 | 38 | 40 | 148
  Asian | 29 | 62 | 36 | 64 | 191
  American Indian or Alaskan Native | 1 | 2 | 0 | 3 | 6
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 2 | 3
  Other | 5 | 0 | 3 | 4 | 12
Number of Migraine Days [Mean (Standard Deviation); unit: days] — A migraine day was defined as when at least 1 of the following situations occurred: A calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours (for CM participants) or at least 2 consecutive hours (for EM participants) of a headache meeting criteria for migraine with or without aura; a calendar day demonstrating at least 4 consecutive hours (for CM participants) or at least 2 consecutive hours (for EM participants) of a headache meeting criteria for probable migraine; a calendar day demonstrating a headache of any duration that was treated with migraine-specific medications.
  days | 13.9 (5.99) | 13.1 (5.49) | 13.6 (5.86) | 13.2 (5.26) | 13.4 (5.63)
Number of Headache Days of Any Severity [Mean (Standard Deviation); unit: days] — Headaches were subjectively rated by participants as mild, moderate or severe. A headache day of any severity for both CM and EM participants was defined as a calendar day (00:00 to 23:59) where the participant (using the electronic headache diary device) reports: a day with headache pain that lasts at least 4 hours with a peak severity of any severity or; a day when the participant used acute migraine-specific medication (triptans or ergots) to treat a headache of any severity or duration.
  days | 13.6 (6.68) | 12.7 (6.20) | 13.2 (6.32) | 12.9 (6.02) | 13.1 (6.29)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Severe AE was defined as inability to carry out usual activities. Treatment-related AEs were defined as AEs with possible, probable, definite, or missing relationship to study drug. Serious AEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Day 0) up to follow-up visit (Day 533)
Population: Safety population included all participants who received at least 1 dose of fremanezumab.
Measure: Count of Participants; unit: Participants
Arm/Group | TEV-48125 225 mg Monthly: New/Placebo Rollover Participants | TEV-48125 225 mg Monthly: Active Rollover Participants | TEV-48125 675 mg Quarterly: New/Placebo Rollover Participants | TEV-48125 675 mg Quarterly: Active Rollover Participants
Number analyzed (Participants) | 418 | 526 | 419 | 525
Participants
  Any AEs | 365 | 456 | 365 | 426
  Severe AEs | 47 | 51 | 45 | 50
  Treatment-related AEs | 263 | 288 | 242 | 270
  Serious AEs | 27 | 29 | 36 | 23
  AEs leading to discontinuation from study | 18 | 18 | 22 | 18

2. Other Pre Specified Outcome: Change From Baseline in Monthly Average Number of Migraine Days During the 4-Week Period at Month 12
Description: A migraine day was defined as when at least 1 of the following situations occurred: A calendar day(0:00 to 23:59) demonstrating at least 4 consecutive hours (for CM participants) or at least 2 consecutive hours (for EM participants) of a headache meeting criteria for migraine with or without aura; a calendar day(0:00 to 23:59) demonstrating at least 4 consecutive hours (for CM participants) or at least 2 consecutive hours (for EM participants) of a headache meeting criteria for probable migraine, a migraine subtype where only 1 migraine criterion was missing; a calendar day(0:00 to 23:59) demonstrating a headache of any duration that was treated with migraine-specific medications (triptans and ergot compounds). Monthly averages were derived and normalized to 28 days equivalent by formula: (number of days of efficacy variable over relevant period/number of days with assessments recorded in e-diary over relevant period)*28. Change was calculated as post-baseline value - baseline value.
Time Frame: Baseline (Day -28 to Day -1), Month 12
Population: Full analysis set (FAS):all participants who received at least 1 dose of fremanezumab, had at least 10 days of efficacy assessments by e-diary after first injection for this study. Data for this outcome was collected and reported separately for CM and EM participants.'Overall number of participants analyzed'=participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: days/month
Groups:
- TEV-48125 225 mg Monthly: New/Placebo Rollover CM Participants: Participants with CM who were randomized to the placebo treatment group or participants who did not rollover from the pivotal efficacy study, received fremanezumab 675 mg SC as loading dose (3 injections of fremanezumab 225 mg/1.5 mL on Day 0) followed by 11 monthly SC doses of fremanezumab at 225 mg (1 injection of fremanezumab 225 mg/1.5mL and 2 injections of placebo 1.5 mL on Days 84, 168, and 252; and 1 injection of fremanezumab 225 mg/1.5mL on Days 28, 56, 112, 140, 196, 224, 280, 308).
- TEV-48125 225 mg Monthly: Active Rollover CM Participants: Participants with CM who were randomized to the active treatment group (Fremanezumab 675/225 mg) in the pivotal efficacy study, received fremanezumab 675 mg SC as loading dose (3 injections of fremanezumab 225 mg/1.5 mL on Day 0) followed by 11 monthly SC doses of fremanezumab at 225 mg (1 injection of fremanezumab 225 mg/1.5mL and 2 injections of placebo 1.5 mL on Days 84, 168, and 252; and 1 injection of fremanezumab 225 mg/1.5mL on Days 28, 56, 112, 140, 196, 224, 280, 308).
- TEV-48125 675mg Quarterly:New/Placebo Rollover CM Participants: Participants with CM who were randomized to the placebo treatment group or participants who did not rollover from the pivotal efficacy study, received fremanezumab 675 mg SC once every 3 months for 12 months for a total of 4 doses (3 injections of fremanezumab 225 mg/1.5mL on Days 0, 84, 168, and 252; and 1 injection of placebo 1.5 mL on Days 28, 56, 112, 140, 196, 224, 280, 308).
- TEV-48125 675 mg Quarterly: Active Rollover CM Participants: Participants with CM who were randomized to the active treatment group (Fremanezumab 675 mg) in the pivotal efficacy study, received fremanezumab 675 mg SC once every 3 months for 12 months for a total of 4 doses (3 injections of fremanezumab 225 mg/1.5mL on Days 0, 84, 168, and 252; and 1 injection of placebo 1.5 mL on Days 28, 56, 112, 140, 196, 224, 280, 308).
- TEV-48125 225 mg Monthly: New/Placebo Rollover EM Participants: Participants with EM who were randomized to the placebo treatment group or participants who did not rollover from the pivotal efficacy study, received 12 monthly SC doses of fremanezumab at 225 mg (1 injection of fremanezumab 225 mg/1.5mL and 2 injections of placebo 1.5 mL on Days 0, 84, 168, and 252; and 1 injection of fremanezumab 225 mg/1.5mL on Days 28, 56, 112, 140, 196, 224, 280, 308).
- TEV-48125 225 mg Monthly: Active Rollover EM Participants: Participants with EM who were randomized to the active treatment group (Fremanezumab 225 mg) in the pivotal efficacy study, received 12 monthly SC doses of fremanezumab at 225 mg (1 injection of fremanezumab 225 mg/1.5mL and 2 injections of placebo 1.5 mL on Days 0, 84, 168, and 252; and 1 injection of fremanezumab 225 mg/1.5mL on Days 28, 56, 112, 140, 196, 224, 280, 308).
- TEV-48125 675mg Quarterly:New/Placebo Rollover EM Participants: Participants with EM who were randomized to the placebo treatment group or participants who did not rollover from the pivotal efficacy study, received fremanezumab 675 mg SC once every 3 months for 12 months for a total of 4 doses (3 injections of fremanezumab 225 mg/1.5mL on Days 0, 84, 168, and 252; and 1 injection of placebo 1.5 mL on Days 28, 56, 112, 140, 196, 224, 280, 308).
- TEV-48125 675 mg Quarterly: Active Rollover EM Participants: Participants with EM who were randomized to the active treatment group (Fremanezumab 675 mg) in the pivotal efficacy study, received fremanezumab 675 mg SC once every 3 months for 12 months for a total of 4 doses (3 injections of fremanezumab 225 mg/1.5mL on Days 0, 84, 168, and 252; and 1 injection of placebo 1.5 mL on Days 28, 56, 112, 140, 196, 224, 280, 308).
Arm/Group | TEV-48125 225 mg Monthly: New/Placebo Rollover CM Participants | TEV-48125 225 mg Monthly: Active Rollover CM Participants | TEV-48125 675mg Quarterly:New/Placebo Rollover CM Participants | TEV-48125 675 mg Quarterly: Active Rollover CM Participants | TEV-48125 225 mg Monthly: New/Placebo Rollover EM Participants | TEV-48125 225 mg Monthly: Active Rollover EM Participants | TEV-48125 675mg Quarterly:New/Placebo Rollover EM Participants | TEV-48125 675 mg Quarterly: Active Rollover EM Participants
Number analyzed (Participants) | 192 | 233 | 194 | 230 | 124 | 173 | 138 | 173
days/month | -7.8 (6.98) | -8.2 (6.14) | -7.6 (6.87) | -7.0 (6.54) | -4.5 (4.20) | -5.5 (4.01) | -5.5 (3.65) | -5.0 (3.78)

3. Other Pre Specified Outcome: Change From Baseline in Monthly Average Number of Headache Days of Any Severity During the 4-Week Period at Month 12
Description: Headaches were subjectively rated by participants as mild, moderate or severe. A headache day of any severity for both CM and EM participants was defined as a calendar day (00:00 to 23:59) where the participant (using the electronic headache diary device) reports: a day with headache pain that lasts at least 4 hours with a peak severity of any severity or; a day when the participant used acute migraine-specific medication (triptans or ergots) to treat a headache of any severity or duration. Monthly averages were derived and normalized to 28 days equivalent by the following formula: (number of days of efficacy variable over relevant period/number of days with assessments recorded in the e-diary over the relevant period) * 28. The change was calculated as post-baseline value - baseline value.
Time Frame: Baseline (Day -28 to Day -1), Month 12
Population: FAS: all participants who received at least 1 dose of fremanezumab, and had at least 10 days of efficacy assessments by electronic diary after first injection for this study. Data for this outcome was collected and reported separately for CM and EM participants. 'Overall number of participants analyzed' = participants evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: days/month
Arm/Group | TEV-48125 225 mg Monthly: New/Placebo Rollover CM Participants | TEV-48125 225 mg Monthly: Active Rollover CM Participants | TEV-48125 675mg Quarterly:New/Placebo Rollover CM Participants | TEV-48125 675 mg Quarterly: Active Rollover CM Participants | TEV-48125 225 mg Monthly: New/Placebo Rollover EM Participants | TEV-48125 225 mg Monthly: Active Rollover EM Participants | TEV-48125 675mg Quarterly:New/Placebo Rollover EM Participants | TEV-48125 675 mg Quarterly: Active Rollover EM Participants
Number analyzed (Participants) | 192 | 233 | 194 | 230 | 124 | 173 | 138 | 173
days/month | -7.7 (6.79) | -7.9 (6.01) | -7.2 (6.48) | -7.1 (6.88) | -4.4 (4.25) | -5.0 (3.90) | -5.0 (3.63) | -4.8 (3.74)

4. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormal Serum Chemistry Results
Description: Potentially clinically significant abnormal serum chemistry findings included: Blood Urea Nitrogen (BUN): greater than or equal to (>=) 10.71 millimoles/liter (mmol/L), creatinine: >=177 micromoles/liter (µmol/L), bilirubin: >=34.2 µmol/L, Alanine Aminotransferase (ALT) (units/liter [U/L]): >=3*upper limit of normal (ULN) Aspartate Aminotransferase (AST) (U/L): >=3*ULN, and Gamma Glutamyl Transferase (GGT) (U/L): >=3*ULN. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Day 0) up to end of treatment (EOT) visit (Day 336)
Population: Safety population included all participants who received at least 1 dose of fremanezumab. Here, 'Overall number of participants analyzed'=participants with both baseline and post-baseline serum chemistry values.
Measure: Count of Participants; unit: Participants
Arm/Group | TEV-48125 225 mg Monthly: New/Placebo Rollover Participants | TEV-48125 225 mg Monthly: Active Rollover Participants | TEV-48125 675 mg Quarterly: New/Placebo Rollover Participants | TEV-48125 675 mg Quarterly: Active Rollover Participants
Number analyzed (Participants) | 408 | 518 | 412 | 513
Participants | 27 | 26 | 11 | 23

5. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormal Hematology Results
Description: Potentially clinically significant abnormal hematology findings included: hemoglobin: less than (<) 115 grams/liter (g/L) (in males) or less than or equal to (<=) 95 g/L (in females), hematocrit: <0.37 L/L (in male) or <0.32 L/L (in female), leukocytes: >=20*10^9/L or <=3*10^9/L, eosinophils/leukocytes: >=10%, and platelets: >=700*10^9/L or <=75*10^9/L. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Day 0) up to EOT visit (Day 336)
Population: Safety population included all participants who received at least 1 dose of fremanezumab. Here, 'Overall number of participants analyzed'=participants with both baseline and post-baseline hematology parameter values.
Measure: Count of Participants; unit: Participants
Arm/Group | TEV-48125 225 mg Monthly: New/Placebo Rollover Participants | TEV-48125 225 mg Monthly: Active Rollover Participants | TEV-48125 675 mg Quarterly: New/Placebo Rollover Participants | TEV-48125 675 mg Quarterly: Active Rollover Participants
Number analyzed (Participants) | 408 | 518 | 412 | 513
Participants | 34 | 39 | 27 | 40

6. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormal Urinalysis Laboratory Tests Results
Description: Potentially clinically significant abnormal urinalysis findings included: blood: >=2 unit increase from baseline, urine glucose (milligrams/decilitre [mg/dL]): >=2 unit increase from baseline, ketones (mg/dL): >=2 unit increase from baseline, urine protein (mg/dL): >=2 unit increase from baseline. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Day 0) up to EOT visit (Day 336)
Population: Safety population included all participants who received at least 1 dose of fremanezumab. Here, 'Overall number of participants analyzed'=participants with both baseline and post-baseline urinalysis values.
Measure: Count of Participants; unit: Participants
Arm/Group | TEV-48125 225 mg Monthly: New/Placebo Rollover Participants | TEV-48125 225 mg Monthly: Active Rollover Participants | TEV-48125 675 mg Quarterly: New/Placebo Rollover Participants | TEV-48125 675 mg Quarterly: Active Rollover Participants
Number analyzed (Participants) | 408 | 517 | 412 | 513
Participants | 128 | 170 | 120 | 146

7. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormal Vital Signs Values
Description: Potentially clinically significant abnormal vital signs findings included: pulse rate: <=50 beats/minute (bpm) and decrease of >=15 bpm, or >=120 bpm and increase of >=15 bpm; systolic blood pressure: <=90 millimeters of mercury (mmHg) and decrease of >=20 mmHg, or >=180 mmHg and increase of >=20 mmHg; diastolic blood pressure: <=50 mmHg and decrease of >=15 mmHg or >=105 mmHg and increase of >=15 mmHg; respiratory rate: <10 breaths/minute; and body temperature >=38.3 degrees centigrade and change of >=1.1 degrees centigrade. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Day 0) up to EOT visit (Day 336)
Population: Safety population included all participants who received at least 1 dose of fremanezumab. Here, 'Overall number of participants analyzed'=participants with both baseline and post-baseline vital signs values.
Measure: Count of Participants; unit: Participants
Arm/Group | TEV-48125 225 mg Monthly: New/Placebo Rollover Participants | TEV-48125 225 mg Monthly: Active Rollover Participants | TEV-48125 675 mg Quarterly: New/Placebo Rollover Participants | TEV-48125 675 mg Quarterly: Active Rollover Participants
Number analyzed (Participants) | 415 | 520 | 414 | 519
Participants | 20 | 33 | 24 | 40

8. Primary Outcome: Number of Participants With Shift From Baseline to Endpoint in Electrocardiogram (ECG) Parameters
Description: ECG parameters included: heart rate, PR interval, QRS interval, QT interval corrected using the Fridericia formula (QTcF), QT interval corrected using the Bazett's formula (QTcB) and RR interval. Shifts represented as Baseline - endpoint value (last observed post-baseline value). Abnormal NCS indicated an abnormal but not clinically significant finding. Abnormal CS indicated an abnormal and clinically significant finding. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Day 0), endpoint (Day 336)
Population: Safety population included all participants who received at least 1 dose of fremanezumab. Here, 'Overall number of participants analyzed' = participants with both baseline and endpoint electrocardiogram findings.
Measure: Count of Participants; unit: Participants
Arm/Group | TEV-48125 225 mg Monthly: New/Placebo Rollover Participants | TEV-48125 225 mg Monthly: Active Rollover Participants | TEV-48125 675 mg Quarterly: New/Placebo Rollover Participants | TEV-48125 675 mg Quarterly: Active Rollover Participants
Number analyzed (Participants) | 386 | 492 | 391 | 489
Participants
  Normal - Normal | 239 | 295 | 230 | 296
  Normal - Abnormal NCS | 45 | 64 | 49 | 67
  Normal - Abnormal CS | 0 | 0 | 0 | 1
  Abnormal NCS - Normal | 42 | 53 | 43 | 60
  Abnormal NCS - Abnormal NCS | 60 | 79 | 69 | 65
  Abnormal NCS - Abnormal CS | 0 | 1 | 0 | 0
  Abnormal CS - Normal | 0 | 0 | 0 | 0
  Abnormal CS - Abnormal NCS | 0 | 0 | 0 | 0
  Abnormal CS - Abnormal CS | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Shift From Baseline to Endpoint in Coagulation Laboratory Test Results
Description: Coagulation parameters included: prothrombin time (PT) (seconds), prothrombin international normalized ratio (INR), activated partial thromboplastin time (aPTT) (seconds). Shifts represented as Baseline - endpoint value (last observed post-baseline value). Shifts from baseline to endpoint were summarized using participant counts grouped into three categories: - Low (below normal range) - Normal (within the normal range of 9.4 to 12.5 seconds) - High (above normal range). A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Day 0), endpoint (Day 336)
Population: Safety population included all participants who received at least 1 dose of fremanezumab. Here, 'Overall number of participants analyzed' = participants with both baseline and endpoint coagulation laboratory test results. 'Number analyzed' = participants evaluable for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | TEV-48125 225 mg Monthly: New/Placebo Rollover Participants | TEV-48125 225 mg Monthly: Active Rollover Participants | TEV-48125 675 mg Quarterly: New/Placebo Rollover Participants | TEV-48125 675 mg Quarterly: Active Rollover Participants
Number analyzed (Participants) | 407 | 516 | 410 | 513
Participants
  PT: Low-Low | 0 | 0 | 0 | 0
  PT: Low-Normal | 1 | 2 | 2 | 1
  PT: Low-High | 0 | 0 | 0 | 0
  PT: Normal-Low | 1 | 3 | 3 | 2
  PT: Normal-Normal | 370 | 465 | 374 | 451
  PT: Normal-High | 10 | 10 | 14 | 14
  PT: High-Low | 0 | 0 | 0 | 0
  PT: High-Normal | 18 | 25 | 9 | 35
  PT: High-High | 7 | 11 | 8 | 10
  Prothrombin INR: number analyzed (Participants) | 406 | 516 | 410 | 513
  Prothrombin INR: Low-Low | 0 | 1 | 4 | 1
  Prothrombin INR: Low-Normal | 11 | 11 | 11 | 9
  Prothrombin INR: Low-High | 0 | 0 | 0 | 0
  Prothrombin INR: Normal-Low | 12 | 15 | 9 | 7
  Prothrombin INR: Normal-Normal | 366 | 468 | 372 | 472
  Prothrombin INR: Normal-High | 6 | 5 | 4 | 4
  Prothrombin INR: High-Low | 0 | 0 | 0 | 1
  Prothrombin INR: High-Normal | 7 | 11 | 6 | 13
  Prothrombin INR: High-High | 4 | 5 | 4 | 6
  aPTT: number analyzed (Participants) | 406 | 516 | 410 | 513
  aPTT: Low-Low | 2 | 2 | 1 | 0
  aPTT: Low-Normal | 4 | 1 | 7 | 7
  aPTT: Low-High | 0 | 1 | 0 | 0
  aPTT: Normal-Low | 3 | 11 | 7 | 10
  aPTT: Normal-Normal | 341 | 423 | 334 | 414
  aPTT: Normal-High | 14 | 18 | 19 | 22
  aPTT: High-Low | 0 | 0 | 0 | 1
  aPTT: High-Normal | 26 | 43 | 26 | 37
  aPTT: High-High | 16 | 17 | 16 | 22

10. Other Pre Specified Outcome: Percentage of Participants With At Least 50% Reduction From Baseline in Monthly Average Number of Migraine Days During the 4-Week Period at Month 12
Description: A migraine day was defined as when at least 1 of the following situations occurred: A calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours (for CM participants) or at least 2 consecutive hours (for EM participants) of a headache meeting criteria for migraine with or without aura; a calendar day (0:00 to 23:59) demonstrating at least 4 consecutive hours (for CM participants) or at least 2 consecutive hours (for EM participants) of a headache meeting criteria for probable migraine, a migraine subtype where only 1 migraine criterion was missing; a calendar day (0:00 to 23:59) demonstrating a headache of any duration that was treated with migraine-specific medications (triptans and ergot compounds). Monthly averages were derived and normalized to 28 days equivalent by formula: (number of days of efficacy variable over relevant period/number of days with assessments recorded in e-diary over relevant period) * 28.
Time Frame: Baseline (Day -28 to Day -1), Month 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | TEV-48125 225 mg Monthly: New/Placebo Rollover CM Participants | TEV-48125 225 mg Monthly: Active Rollover CM Participants | TEV-48125 675mg Quarterly:New/Placebo Rollover CM Participants | TEV-48125 675 mg Quarterly: Active Rollover CM Participants | TEV-48125 225 mg Monthly: New/Placebo Rollover EM Participants | TEV-48125 225 mg Monthly: Active Rollover EM Participants | TEV-48125 675mg Quarterly:New/Placebo Rollover EM Participants | TEV-48125 675 mg Quarterly: Active Rollover EM Participants
Number analyzed (Participants) | 195 | 240 | 197 | 237 | 125 | 174 | 139 | 174
percentage of participants | 54 | 59 | 52 | 54 | 58 | 75 | 68 | 64

11. Other Pre Specified Outcome: Percentage of Participants With At Least 50% Reduction From Baseline in Monthly Average Number of Headache Days of at Least Moderate Severity During the 4-Week Period
Description: Headaches were subjectively rated by participants as mild, moderate or severe. A headache day of at least moderate severity for both CM and EM participants was defined as a calendar day (00:00 to 23:59) where the participant (using the electronic headache diary device) reports: a day with headache pain that lasts at least 4 hours with a peak severity of at least moderate severity or; a day when the participant used acute migraine-specific medication (triptans or ergots) to treat a headache of any severity or duration. Monthly averages were derived and normalized to 28 days equivalent by the following formula: (number of days of efficacy variable over relevant period/number of days with assessments recorded in the e-diary over the relevant period) * 28.
Time Frame: Baseline (Day -28 to Day -1), Month 12
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | TEV-48125 225 mg Monthly: New/Placebo Rollover CM Participants | TEV-48125 225 mg Monthly: Active Rollover CM Participants | TEV-48125 675mg Quarterly:New/Placebo Rollover CM Participants | TEV-48125 675 mg Quarterly: Active Rollover CM Participants | TEV-48125 225 mg Monthly: New/Placebo Rollover EM Participants | TEV-48125 225 mg Monthly: Active Rollover EM Participants | TEV-48125 675mg Quarterly:New/Placebo Rollover EM Participants | TEV-48125 675 mg Quarterly: Active Rollover EM Participants
Number analyzed (Participants) | 193 | 240 | 197 | 237 | 124 | 174 | 138 | 174
percentage of participants | 56 | 62 | 54 | 54 | 58 | 72 | 67 | 68

12. Primary Outcome: Number of Participants With Injection Site Reactions
Description: Number of participants who reported treatment-emergent injection site reactions are summarized. Preferred terms from MedDRA version 18.1 were offered without a threshold applied. Injection site reactions included injection site induration, pain, erythema, haemorrhage, pruritus, swelling, bruising, rash, urticaria, warmth, dermatitis, haematoma, inflammation, discolouration, discomfort, hypersensitivity, hypoaesthesia, irritation, oedema, papule, paraesthesia, vesicles and pallor. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline (Day -28 to Day -1), Month 12
Population: Safety population included all participants who received at least 1 dose of fremanezumab.
Measure: Count of Participants; unit: Participants
Arm/Group | TEV-48125 225 mg Monthly: New/Placebo Rollover Participants | TEV-48125 225 mg Monthly: Active Rollover Participants | TEV-48125 675 mg Quarterly: New/Placebo Rollover Participants | TEV-48125 675 mg Quarterly: Active Rollover Participants
Number analyzed (Participants) | 418 | 526 | 419 | 525
Participants
  Injection site induration | 167 | 174 | 144 | 134
  Injection site pain | 149 | 156 | 135 | 140
  Injection site erythema | 130 | 144 | 99 | 124
  Injection site haemorrhage | 34 | 38 | 21 | 38
  Injection site pruritus | 31 | 43 | 17 | 24
  Injection site swelling | 7 | 10 | 6 | 8
  Injection site bruising | 2 | 2 | 4 | 3
  Injection site rash | 4 | 2 | 5 | 2
  Injection site urticaria | 4 | 2 | 3 | 2
  Injection site warmth | 3 | 2 | 1 | 1
  Injection site dermatitis | 0 | 1 | 0 | 1
  Injection site haematoma | 1 | 0 | 0 | 1
  Injection site inflammation | 0 | 1 | 1 | 0
  Injection site discolouration | 0 | 1 | 0 | 0
  Injection site discomfort | 0 | 0 | 0 | 1
  Injection site hypersensitivity | 1 | 0 | 0 | 0
  Injection site hypoaesthesia | 1 | 1 | 0 | 0
  Injection site irritation | 0 | 0 | 0 | 1
  Injection site oedema | 1 | 1 | 1 | 0
  Injection site papule | 1 | 0 | 0 | 0
  Injection site paraesthesia | 0 | 0 | 1 | 0
  Injection site vesicles | 0 | 1 | 1 | 0
  Injection site pallor | 0 | 0 | 0 | 1

13. Primary Outcome: Number of Participants With Suicidal Ideation and Suicidal Behavior as Assessed by the Electronic Columbia-Suicide Severity Rating Scale (eC-SSRS)
Description: eC-SSRS is a questionnaire to assess suicidal ideation and suicidal behavior. Suicidal behavior was defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation was defined as a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent, any self-injurious behavior with no suicidal intent.
Time Frame: Baseline (Day -28 to Day -1), Month 12
Population: Safety population included all participants who received at least 1 dose of fremanezumab.
Measure: Count of Participants; unit: Participants
Arm/Group | TEV-48125 225 mg Monthly: New/Placebo Rollover Participants | TEV-48125 225 mg Monthly: Active Rollover Participants | TEV-48125 675 mg Quarterly: New/Placebo Rollover Participants | TEV-48125 675 mg Quarterly: Active Rollover Participants
Number analyzed (Participants) | 418 | 526 | 419 | 525
Participants
  Suicidal ideation | 2 | 0 | 2 | 1
  Suicidal attempt | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day 0) up to follow-up visit (Day 533)
Description: Safety population included all participants who received at least 1 dose of fremanezumab.
Arm/Group | TEV-48125 225 mg Monthly: New/Placebo Rollover Participants | TEV-48125 225 mg Monthly: Active Rollover Participants | TEV-48125 675 mg Quarterly: New/Placebo Rollover Participants | TEV-48125 675 mg Quarterly: Active Rollover Participants
All-Cause Mortality (participants affected / at risk) | 0/418 | 0/526 | 1/419 | 0/525
Serious Adverse Events (participants affected / at risk) | 27/418 | 29/526 | 36/419 | 23/525
Other Adverse Events (participants affected / at risk) | 300/418 | 367/526 | 284/419 | 329/525
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | TEV-48125 225 mg Monthly: New/Placebo Rollover Participants (N=418) | TEV-48125 225 mg Monthly: Active Rollover Participants (N=526) | TEV-48125 675 mg Quarterly: New/Placebo Rollover Participants (N=419) | TEV-48125 675 mg Quarterly: Active Rollover Participants (N=525)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Congenital cystic disease of liver (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hereditary haemochromatosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petrositis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ammonia increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/365 (0) | 0/454 (0) | 1/369 (1) | 0/457 (0) — This is a gender-specific AE. Only female participants were at risk.
High grade B-cell lymphoma Burkitt-like lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Phyllodes tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/54 (0) | 0/72 (0) | 1/51 (1) | 0/68 (0) — This is a gender-specific AE. Only male participants were at risk.
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cluster headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Perineurial cyst (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Primary progressive multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Status migrainosus (Nervous system disorders) | 2 (4) | 1 (1) | 1 (1) | 0 (0)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/365 (0) | 1/454 (1) | 0/369 (0) | 0/457 (0) — This is a gender-specific AE. Only female participants were at risk.
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0/365 (0) | 1/454 (1) | 0/369 (0) | 0/457 (0) — This is a gender-specific AE. Only female participants were at risk.
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1/365 (1) | 0/454 (0) | 0/369 (0) | 0/457 (0) — This is a gender-specific AE. Only female participants were at risk.
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0/365 (0) | 0/454 (0) | 1/369 (1) | 0/457 (0) — This is a gender-specific AE. Only female participants were at risk.
Adjustment disorder with mixed disturbance of emotion and conduct (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1/365 (1) | 0/454 (0) | 0/369 (0) | 0/457 (0) — This is a gender-specific AE. Only female participants were at risk.
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0/365 (0) | 1/454 (1) | 0/369 (0) | 0/457 (0) — This is a gender-specific AE. Only female participants were at risk.
Ovarian cyst (Reproductive system and breast disorders) | 1/365 (1) | 0/454 (0) | 0/369 (0) | 0/457 (0) — This is a gender-specific AE. Only female participants were at risk.
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1/365 (1) | 0/454 (0) | 0/369 (0) | 1/457 (1) — This is a gender-specific AE. Only female participants were at risk.
Ovarian mass (Reproductive system and breast disorders) | 1/365 (1) | 0/454 (0) | 0/369 (0) | 0/457 (0) — This is a gender-specific AE. Only female participants were at risk.
Uterine haemorrhage (Reproductive system and breast disorders) | 1/365 (1) | 0/457 (0) | 0/369 (0) | 0/457 (0) — This is a gender-specific AE. Only female participants were at risk.
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salpingo-oophorectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TEV-48125 225 mg Monthly: New/Placebo Rollover Participants (N=418) | TEV-48125 225 mg Monthly: Active Rollover Participants (N=526) | TEV-48125 675 mg Quarterly: New/Placebo Rollover Participants (N=419) | TEV-48125 675 mg Quarterly: Active Rollover Participants (N=525)
Injection site erythema (General disorders) | 130 (430) | 144 (446) | 99 (284) | 124 (386)
Injection site haemorrhage (General disorders) | 34 (43) | 38 (66) | 21 (38) | 38 (62)
Injection site induration (General disorders) | 167 (717) | 174 (753) | 144 (543) | 134 (666)
Injection site pain (General disorders) | 149 (980) | 156 (982) | 135 (981) | 140 (811)
Injection site pruritus (General disorders) | 31 (101) | 43 (107) | 17 (64) | 24 (64)
Bronchitis (Infections and infestations) | 24 (25) | 15 (16) | 20 (22) | 24 (26)
Influenza (Infections and infestations) | 14 (18) | 27 (29) | 8 (9) | 25 (28)
Nasopharyngitis (Infections and infestations) | 43 (61) | 69 (107) | 37 (58) | 68 (108)
Sinusitis (Infections and infestations) | 30 (40) | 27 (28) | 28 (35) | 31 (38)
Upper respiratory tract infection (Infections and infestations) | 55 (65) | 62 (76) | 73 (97) | 63 (78)
Urinary tract infection (Infections and infestations) | 25 (38) | 27 (43) | 26 (29) | 33 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2016-03-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT02638103/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT02638103/SAP_001.pdf